CLINICAL TRIAL: NCT01104636
Title: "VIBRATIONS": Varenicline In Patients Ambitioned To Terminate Smoking - A Non-Interventional Study
Brief Title: "VIBRATIONS" - A Study In Smokers Who Are Willing And Motivated To Stop Smoking With The Aid Of Varenicline Which Will Be Prescribed According To Usual Clinical Practice In Germany
Acronym: VIBRATIONS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051141
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group prospective treatment cohort (varenicline)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — varenicline tablets prescribed as per local German SmPC for 12 weeks duration

SUMMARY:
The aim of this study is to determine the success rates for stopping smoking with varenicline in Germany. The main measure of success will be continuous abstinence from smoking (not a single puff) in the last week of the standard 12 week treatment period. Additional information will be gathered regarding prescribing practices in Germany, smoking history, reasons why smokers quit smoking and re-start smoking, smoking related illnesses and the tolerability of varenicline.

DETAILED DESCRIPTION:
Sampling Method Details: Non-interventional study: subjects to be selected according to the usual clinical practice of their physician.

ELIGIBILITY:
Inclusion Criteria:

* Legal adult age
* Regular smoker, with main tobacco product smoked being cigarettes, and willing and motivated to stop smoking
* Evidence of a personally signed and dated Informed Consent document.

Exclusion Criteria:

* Any subjects considered unsuitable according to the Summary of product characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult smokers who are willing and motivated to stop smoking
Sampling Method: Non-Probability Sample
Enrollment: 1177 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051141&StudyName=%22VIBRATIONS%22%20-%20A%20Study%20In%20Smokers%20Who%20Are%20Willing%20And%20Motivated%20To%20Stop%20Smoking%20With%20The%20Aid%20Of%20Varenicline%20Which%20Will%20Be%20Pres

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1391 participants were screened and 1177 participants were assigned to the treatment.
Groups:
- Varenicline: Varenicline tartrate tablet was prescribed for 12 weeks as per the approved Summary of Product Characteristics (SmPC) and was adjusted according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Varenicline
Started | 1177
Completed | 999
Not Completed | 178
Not completed — Lack of Efficacy | 43
Not completed — Lost to Follow-up | 24
Not completed — Withdrawal by Subject | 4
Not completed — Other | 43
Not completed — Study terminated by sponsor | 1
Not completed — Pregnancy | 2
Not completed — Adverse Event | 40
Not completed — Ongoing | 21

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 1173
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data for 4 participants was not available.
  years | 49.4 (12.0)
Sex/Gender, Customized [Number; unit: participants] — Demographic data for 4 participants was not available.
  participants
    Male | 669
    Female | 503
    Unspecified | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Abstained From Smoking at Week 12
Description: The use of nicotine was recorded using Nicotine Use Inventory (NUI) to determine the participants who abstained from smoking for the previous 7 days. A responder for the 7-day point prevalence was defined as those with 'no' answers to the following two questions: Did the participant smoke any cigarettes (even a puff) in the last 7 days; and did participant use any other tobacco products (example pipe, cigars, snuff, chewing tobacco) in the last 7 days.
Time Frame: Week 12
Population: The all participants' population included all enrolled participants who had received at least 1 dose (including partial doses) of study medication. Missing observations were not imputed and hence the participants analyzed are the ones without missing values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1035
percentage of participants | 71.1 [68.5 to 73.7]

2. Secondary Outcome: Level of Nicotine Dependence Measured by the Fagerstrom Test
Description: Fagerstrom Test for Nicotine Dependence (FTND) was designed to provide measure of nicotine dependence related to cigarette smoking. It contains 4 yes-no and 2 multiple choice questions. Items are scored 0-3 for multiple choice items, items are summed to yield total score of 0-10 (0=minimum to 10=maximum nicotine dependence).
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Scores on a scale
Arm/Group | Varenicline
Number analyzed (Participants) | 1030
Scores on a scale | 5.30 (2.31)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 7/1177
Other Adverse Events (participants affected / at risk) | 40/1177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1177)
Nausea (Gastrointestinal disorders) | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 2
Apathy (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1177)
Nausea (Gastrointestinal disorders) | 40

LIMITATIONS AND CAVEATS:
It is highly likely that Adverse Events were under reported for this study as it was a Non Interventional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.